CLINICAL TRIAL: NCT03888794
Title: Magnetic Resonance Imaging Versus Four Dimensional Ultrasound in Detection of Central Nervous System Fetal Congenital Anomalies
Brief Title: MRI Versus Four Dimensional Ultrasound in Detection of CNS Fetal Congenital Anomalies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nehal Kamal Mohamed, principal Investigator, Assiut University
Other Study IDs: MRIUSCNS
Record Dates: First submitted 2019-03-19; First posted 2019-03-25 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Congenital Anomalies
MeSH Terms: conditions — Congenital Abnormalities | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Magnetic Resonance Imaging — Magnetic Resonance Imaging on pregnant women after 18 weeks of pregnancy with US diagnosis of congenital CNS fetal abnormality.

SUMMARY:
Congenital central nervous system (CNS) anomalies are common and most devastating. They occur in frequency of about 1.4 to 1.6 per 1000 live births but are seen in about 3-6% of still births.They account for 40% of deaths of all infants in the first year of life. In survivors, they cause a variety of neurological disorders, mental retardation or drug resistant epilepsy.

CNS anomalies are usually compatible with life, prolonged hospitalization, higher health care costs, uncertain future life quality and significant burden to families and society.

DETAILED DESCRIPTION:
Early detection of congenital CNS anomalies gives time available for the clinician and parents to plan about the outcome of pregnancy.

Prenatal ultrasound has been well established for decades as the primary technique for evaluating the developing fetus in normal as well as in high risk cases. Advantages of US include widespread availability, relatively low cost and quick, lack of harmful effect to fetus or mother and real time imaging.

Although ultrasound can characterize many anomalies accurately, it has many limitations as operator dependent, small field of view, and relatively poor soft-tissue contrast, beam attenuation by maternal adipose tissue and fetal bone, limited visualization of posterior fossa after 33 weeks gestation because of calvarial calcification. Also, ultrasound relies heavily on fetal positioning and presence of sufficient amniotic fluid to provide an adequate acoustic window fetus So, US findings are occasionally incomplete or inconclusive to guide treatment choices.

Fetal brain MRI became embraced as a clinically important imaging technique useful for fetal assessment, which is helpful in formulating prognosis and perinatal management and can detect occult abnormalities in up to 50% of cases for certain indications.

It can overcome many of ultrasound limitations as it is not limited by maternal obesity, fetal position, or oligohydramnios. Additionally, it has better soft tissue contrast resolution, as well as the ability to distinguish individual fetal structures such as brain, lung, liver, kidney, and bowel. In addition, visualization of the brain is not restricted by the ossified skull. Moreover, MRI provides multiplanar imaging as well a larger field of view, facilitating examination of fetuses with large or complex anomalies.

ELIGIBILITY:
Inclusion Criteria:

1. All pregnancies with either suspected or detected fetal anomalies on ultrasound excluding first trimester pregnancies (to allow completion of period of organogenesis).
2. Pregnant females with past or family history of congenital fetal abnormality.

Exclusion Criteria:

1. Pregnancies with normal antenatal US.
2. pregnancies in first trimester
3. Claustrophobic patients.
4. contraindication to MRI as cochlear implants and pacemakers.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pregnant females referred from obstetric department with either suspected or detected fetal anomalies on ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-05-20 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Ventricular size | baseline
  assess the ventricular size by measuring the anteroposterior diameter of the fourth ventricle, the width of the third ventricle, and the transverse diameter of the lateral ventricles on the coronal images.

SECONDARY OUTCOMES:
Correlate MRI findings with Ultrasound findings. | baseline
  to correlate fetal biometry and ventricular size with ultrasound findings.

CONTACTS AND LOCATIONS:
Overall Officials: Nehal Mohamed, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Onkar D, Onkar P, Mitra K. Evaluation of Fetal Central Nervous System Anomalies by Ultrasound and Its Anatomical Co-relation. J Clin Diagn Res. 2014 Jun;8(6):AC05-7. doi: 10.7860/JCDR/2014/8052.4437. Epub 2014 Jun 20. PMID 25120962
- [Result] Manganaro L, Bernardo S, Antonelli A, Vinci V, Saldari M, Catalano C. Fetal MRI of the central nervous system: State-of-the-art. Eur J Radiol. 2017 Aug;93:273-283. doi: 10.1016/j.ejrad.2017.06.004. Epub 2017 Jun 17. PMID 28668426
- [Result] Sefidbakht S, Dehghani S, Safari M, Vafaei H, Kasraeian M. Fetal Central Nervous System Anomalies Detected by Magnetic Resonance Imaging: A Two-Year Experience. Iran J Pediatr. 2016 Jun 6;26(4):e4589. doi: 10.5812/ijp.4589. eCollection 2016 Aug. PMID 27729957